CLINICAL TRIAL: NCT05293587
Title: Physical Activity to Reduce Diabetes Risk in Serious Mental Illness: PARCS Pilot Study
Brief Title: Physical Activity to Reduce Diabetes Risk in Serious Mental Illness
Acronym: PARCS Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Vanderbilt University School of Medicine (Other); Kansas State University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Catherine Davis, Professor of Medicine, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1434186; 3P30DK020593-42S1 (NIH); VUMC86160 (Other Grant/Funding Number: Vanderbilt Diabetes Res. & Trng Ctr Pilot/Feasibility Grant)
Record Dates: First submitted 2021-08-18; First posted 2022-03-24 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Mental Disorders, Severe
MeSH Terms: conditions — Mental Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Waitlist control group
Who Masked: Outcomes Assessor
Masking Description: Fitbit data will be analyzed by Kansas State University personnel masked to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): Physical activity sessions at public parks led by a Serenity Behavioral Health Certified Peer Specialist
  Interventions: Behavioral: Physical Activity
- Waitlist (No Intervention): Participants will continue their usual care in the PEERS program. They will be offered the intervention after they have completed posttest measures.

INTERVENTIONS:
Behavioral: Physical Activity — Physical activity sessions will take place 3x/week over six weeks and will take between 45 and 60 minutes for each session. The sessions will be led by a Serenity Behavioral Health CPS as part of the PEERS program and will be supervised by research staff. Sessions will occur at public parks. Transportation to the park will be provided by Serenity Behavioral Health. Structured activities will include a warm-up, a mix of simple exercises requiring minimal supplies (such as walking, basic aerobic movements, and body weight resistance exercises), and cool-down. Sessions will be held in green park environments with shade, restrooms, and level walking paths.
  Other Names: Park-based Physical Activity
  Arms: Physical Activity

SUMMARY:
The aim of this project is to trial the protocol of a park-based physical activity (PA) intervention in adults with severe mental illness (SMI) in a community mental health center's peer support program.

DETAILED DESCRIPTION:
Aim 1: Test the feasibility and acceptability of a park-based PA intervention led by Certified Peer Specialists (CPS) and adapted for adults with SMI. Rationale: Park-based interventions led by CPSs represent a novel approach to increase program satisfaction and adherence to PA behavior change in persons with SMI. Hypothesis 1A: Most (80%) people offered the intervention will participate most of the time (≥2 day/week). Hypothesis 1B: CPSs and SMI patients will express satisfaction with the program (6 on an 8-point scale). Aim 2: Test the effectiveness of a park-based PA intervention led by CPSs on increasing PA and improving fitness in adults with SMI. Rationale: Park-based PA is associated with greater intensity and duration of PA, better fitness, and less obesity and depression, issues that are especially problematic for adults with SMI. Hypothesis 2A: People enrolled in the intervention will engage in more PA than at baseline (90min moderate to vigorous PA (MVPA)/week). Hypothesis 2B: The intervention will result in improved fitness (6 min walk test) relative to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Authorized for peer group treatment through the Serenity behavioral health facility
* Medically cleared for participation
* Able to act as their own legal guardian

Exclusion Criteria:

* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Percent attendance | During 6-week intervention period
  Feasibility will be assessed by attendance to park PA sessions (0-100%). Higher attendance indicates greater engagement with the intervention.
Participant satisfaction | 8 weeks
  Acceptability will be assessed via participant satisfaction, measured using an abbreviated version of the Physical Activity Class Satisfaction Questionnaire (PACSQ). PACSQ is a valid measure for capturing client satisfaction within exercise classes in the following nine dimensions: mastery experiences, cognitive development, teaching, normative success, interaction with others, fun and enjoyment, improvement of health and fitness, diversionary experiences, and relaxation. Each of the dimensions of satisfaction is measured using an 8-point Likert scale, with responses ranging from 1="No satisfaction" to 8="Very satisfying". PACSQ has shown acceptable reliability in each of its subscales (all α's ≥ .85), and survey items are highly correlated with participants' intentions to attend a similar course in the future.

SECONDARY OUTCOMES:
Change in Physical Activity | Baseline, during 6-week intervention period
  Fitbit min/week moderate to vigorous physical activity. Greater min/week physical activity is better.
Change in Aerobic Fitness from Baseline at 8 weeks | Baseline, 8 weeks
  6-minute walk test. Greater distance indicates better fitness.

OTHER OUTCOMES:
Structured Assessment of FEeasibility | Approximately 1 year
  The Structured Assessment of FEeasibility (SAFE) standardized measure will be used to determine overall intervention feasibility. The SAFE measure specifically evaluates interventions within a mental health services framework and includes 16 items that capture information in three categories: intervention, resource consequences, and evaluation. The PI in collaboration with CPSs will complete the SAFE measure. The SAFE measure has demonstrated excellent inter-rater and test-retest reliability (0.84, 95% confidence interval (CI) 0.79-0.89; 0.89, 95% CI 0.85-0.93 respectively). Rather than using a summary score, the individual items should be considered (e.g., yes, partial, no, unable to rate).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Davis, PhD, Principal Investigator — Augusta University; Gina M Besenyi, MPH PhD, Principal Investigator — Kansas State University
Locations (2):
- United States (2):
  - Serenity Behavioral Health System, Augusta, Georgia
  - Georgia Prevention Institute, Augusta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with colleagues who have a reasonable request and analysis plan with appropriate credit.
Supporting Information: Study Protocol, ICF